CLINICAL TRIAL: NCT02354729
Title: Using Text Messaging and Financial Incentives to Encourage Allergic Young Adults to Carry Epinephrine
Brief Title: Encouraging Allergic Young Adults to Carry Epinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carolyn Cannuscio, Assistant Professor of Family Medicine and Community Health, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UPenn
Record Dates: First submitted 2015-01-23; First posted 2015-02-03 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Adherence; Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Economics, Behavioral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants received text messages and financial incentives after successfully documenting that they were carrying their epinephrine auto-injectors, based on principles of behavioral economics.
  Interventions: Other: Behavioral Economics
- Control (No Intervention): Participants received text messages.

INTERVENTIONS:
Other: Behavioral Economics — Use financial incentives to promote epinephrine-carrying.
  Arms: Intervention

SUMMARY:
Fifteen million Americans suffer from food allergies. Food allergies can be life threatening; the only known life-saving treatment is epinephrine. Adolescents/young adults are at increased risk of adverse events, because of increased risk-taking with food and decreased likelihood of carrying epinephrine. This is a pilot randomized trial to test text message reminders, with and without financial incentives, to encourage allergic young adults to carry epinephrine.

DETAILED DESCRIPTION:
Aim: We pilot tested a novel strategy to encourage young adults with food allergies to carry their epinephrine auto-injectors. Adolescents/young adults are at increased risk of adverse events, because of increased risk-taking with food and decreased likelihood of carrying epinephrine.

Study design: This is a pilot randomized controlled trial, with a survey component. Text messaging is the mode of communication and inquiry with study participants.

Hypothesis: The intervention group, which will receive modest financial incentives for carrying epinephrine, will be more likely to demonstrate that they are carrying their epinephrine, when queried by the study team.

This study employs text messaging, along with photography, as a mode of momentary ecologic assessment, or real-time measurement of epinephrine carrying. In addition, text messaging was used as a mode of asking questions regarding food allergy knowledge and beliefs among young adults. Text messages were sent from a designated telephone (and telephone number) purchased for use in this study. We used text messaging for reminder messages, text responses, and for the participants to send photographs back to us. We converted text message data (participants responses) into a RedCap database. Our research coordinator sent and received the text messages and compiled a secure RedCap database of responses.

ELIGIBILITY:
Inclusion Criteria:

* Have known food allergy
* Epinephrine auto-injector prescription
* Access to a cell phone with ability to send picture messages

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Proportion of check-ins at which participant is carrying epinephrine | 10 randomly timed check-ins during the 7 week intervention period
  Proportion of check-ins at which participants were successfully carrying their epinephrine, measured using cell phone photographs.

SECONDARY OUTCOMES:
Self-reported acceptability of text messages | Measured at the end of the 7 week intervention
  Assess young adults' perspectives on text messaging as a vehicle for communicating health messages.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn C Cannuscio, ScD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Result] Cannuscio CC, Dupuis R, Graves A, Seymour JW, Kounaves S, Strupp E, Leri D, Frasso R, Grande D, Meisel ZF. A behavioral economics intervention to encourage epinephrine-carrying among food-allergic adults: a randomized controlled trial. Ann Allergy Asthma Immunol. 2015 Sep;115(3):234-240.e1. doi: 10.1016/j.anai.2015.05.018. Epub 2015 Jun 17. PMID 26093776